CLINICAL TRIAL: NCT00003308
Title: A Phase II Trial of Radiosurgery for 1 to 3 Newly Diagnosed Brain Metastases From Renal Cell, Melanoma and Sarcoma
Brief Title: Radiation Therapy in Treating Patients With Newly Diagnosed Brain Metastases From Kidney Cancer, Melanoma, or Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066255; E-6397
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Kidney Cancer; Melanoma (Skin); Metastatic Cancer; Ovarian Cancer; Sarcoma
Keywords: metastatic osteosarcoma; chondrosarcoma; stage IV renal cell cancer; stage IV melanoma; tumors metastatic to brain; stage IV uterine sarcoma; ovarian sarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Neoplasm Metastasis; Ovarian Neoplasms; Sarcoma; Osteosarcoma; Chondrosarcoma; Carcinoma, Renal Cell; Brain Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Radiosurgery

INTERVENTIONS:
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy in treating patients with newly diagnosed brain metastases from kidney cancer, melanoma, or sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate whether the delivery of stereotactic radiosurgery without conventional whole brain radiotherapy is feasible in patients with 1-3 newly diagnosed brain metastases from renal cell carcinoma, melanoma, or sarcoma.
* Determine the 3-, 6-, and 12-month radiographic and neurologic intracranial patterns of progression (i.e., original lesions vs new lesions) in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to maximum tumor diameter (2 cm vs greater than 2 cm to 3 cm vs greater than 3 cm to 4 cm).

Patients undergo stereotactic radiosurgery at an assigned dose according to tumor diameter. Patients undergo MRI or CT scan at 3, 6, and 12 months after treatment or until disease progression.

All other therapies are allowed after stereotactic radiosurgery except external beam whole brain radiotherapy or resection of brain metastases, unless there is documented progression or unrelenting mass effect that necessitates craniotomy.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 7.2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma, melanoma, or sarcoma with 1-3 newly diagnosed intraparenchymal brain metastases based on contrast-enhanced MRI (CT scan acceptable if patients have a medical contraindication to MRI)
* No lesion greater than 4.0 cm in diameter and, if multiple lesions are present, no more than one greater than 3.0 cm in diameter
* No limitation on the extent of extracranial metastatic disease
* No metastases in the brain stem, midbrain, pons, or medulla
* No leptomeningeal metastases documented by MRI or CSF evaluation
* No metastases within 10 mm of optic nerve or chiasm
* No history of multiple liver metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 50,000/mm^3
* Hemoglobin greater than 8 g/dL

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No major medical illness
* No psychoses
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy allowed
* Systemic chemotherapy may be continued at the discretion of investigator after completion of radiosurgery

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior cranial radiotherapy
* Prior or concurrent radiotherapy to noncranial sites allowed

Surgery:

* No prior surgical resection for brain metastases
* Prior stereotactic biopsy for diagnostic purposes allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02-02 (Actual); Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minesh P. Mehta, MD, Study Chair — University of Wisconsin, Madison
Locations (14):
- United States (11):
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Alegent Health-Midlands Community Hospital, Papillion, Nebraska
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Ireland Cancer Center, Cleveland, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Manon R, O'Neill A, Knisely J, Werner-Wasik M, Lazarus HM, Wagner H, Gilbert M, Mehta M; Eastern Cooperative Oncology Group. Phase II trial of radiosurgery for one to three newly diagnosed brain metastases from renal cell carcinoma, melanoma, and sarcoma: an Eastern Cooperative Oncology Group study (E 6397). J Clin Oncol. 2005 Dec 1;23(34):8870-6. doi: 10.1200/JCO.2005.01.8747. PMID 16314647